CLINICAL TRIAL: NCT03729531
Title: The Clinical Effect of No-touch Vein Harvesting Technique in Off-pump Coronary Artery Bypass Graft
Brief Title: Clinical Effect of No-touch Harvesting Technique in OPCABG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Zheng Ju-bing, Clinical investigator, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PX2018027
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Coronary Artery Disease; Graft Failure
Keywords: Coronary Artery Disease; Coronary Artery Bypass Grafting; Vein Graft Failure; Endothelial dysfunction
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): The perivascular tissue is stripped off when harvesting the vein, and saline will be used to distend the vein to check for leakage.
  Interventions: Procedure: Conventional vein harvesting technique
- No-touch (Experimental): The vein will be harvested by frequency electrotome and the perivascular tissue will be preserved, the vein will not be distended.
  Interventions: Procedure: no-touch vein harvesting technique

INTERVENTIONS:
Procedure: Conventional vein harvesting technique — Long incision will be used to expose the vein, the perivascular tissue will be dissected carefully by scissors, to check for leakage, the vein will be distended by injecting saline.
  Arms: Conventional
Procedure: no-touch vein harvesting technique — The vein will be harvested by low-frequency electrotome, about 5mm surrounding tissue will be preserved with the vein, distention should be avoided, the vein will not be cut off until being anastomosed.
  Arms: No-touch

SUMMARY:
This study aims to investigate the clinical effect of the new saphenous vein harvesting technique "No-touch" in off-pump coronary artery bypass grafting(OPCABG), comparing to the conventional technique. Adopting CTA to evaluate the 3 months patency of the graft, we will compare veins harvested using No-touch technique to saphenous veins using conventional open technique.

DETAILED DESCRIPTION:
Coronary artery disease(CAD) is a widespread health issue around the world. It is proven that atherosclerosis is a inflammatory disease, and endothelial dysfunction is one of the key factors that initiates the inflammatory response. Accumulating studies indicate that endothelial homeostasis plays a primordial role in the development of atherosclerosis.

Coronary artery bypass grafting(CABG) is the standard treatment of three-vessel or left main coronary artery disease, and its long-term benefits is apparent. Saphenous vein is the most common graft in CABG, however, the long-term patency is only about 50% in one year, as a result, it is urgent to discover a solution to improve the long term potency of vein grafts.

Conventional harvesting technique dissects the perivascular tissue and inject saline to check leakage, which causes damages to the endothelium of the vein, initiating inflammatory response. No-touch technique is a atraumatic, non-distended harvesting technique. According to the criteria, we will randomize the patients into two groups, the conventional and No-touch group, the vein will be used in sequential anastomosis, by comparing the 3 months patency rate assessed by CTA, we aim to compare the clinical outcomes of the two different vein harvesting techniques.

ELIGIBILITY:
Inclusion Criteria:

* patients from northern China
* first time isolated off-pump coronary artery bypass graft
* echocardiogram show that ejection fraction is over 35%
* the diameter of saphenous vein ≥ 2mm
* the vein graft will be used in sequential anastomosis, and the anastomosis sites ≥2
* be able to sign informed consent form

Exclusion Criteria:

* patients who need to undergo urgent surgery
* Severe renal insufficiency(creatinine >200 umol/L)
* allergic to radiocontrast agent
* vein is used to isolated anastomosis
* Combined with malignant tumor or other severe systemic conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-12-21 (Actual); Primary Completion 2021-06-08 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
short-term patency rate of vein grafts | 3 months after surgery
  the patency of vein grafts will be assessed by CTA, the doctors of CT department will be masked, at least 2 doctors will provide their conclusions.when the results is controversial, the third doctor will be asked to review the image and provide another conclusion, the patency will be assessed according all results.

SECONDARY OUTCOMES:
long-term patency rate of vein grafts | 12 months after surgery
  the patency will be assessed by CTA the same as short-term patency
major adverse cardiac and cerebrovascular events(MACCE) rate | 3 months and 12 months after surgery
  all-cause death, myocardial infarction, stroke,repeat revascularizaiton
CCS grade | 3 months and 12 months after surgery
  the grade of angina wii be assessed according to Canadian Cardiovascular Society standard
the healing of the lower leg incision | 3 months and 12 months after surgery
  the healing of the incision will be divided into primary healing, e.g. less tissue defects, neat wound edges, no infection, adhesion or suture to create a tight wound; delayed healing, which means the wound does not closed within 1 month; infection, the wound does not close after 3 months, or necrotic tissues are seen in the incision.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-bing Zheng, M.D., Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Capital medical university, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peng Z, Zhao R, Yang Y, Hua K, Yang X. Predictive Value of the CT-Based Visceral Adiposity Tissue Index and Triglyceride-Glucose Index on New-Onset Atrial Fibrillation after Off-Pump Coronary Artery Bypass Graft: Analyses from a Longitudinal Study. Rev Cardiovasc Med. 2023 Nov 30;24(11):338. doi: 10.31083/j.rcm2411338. eCollection 2023 Nov. PMID 39076438